CLINICAL TRIAL: NCT00801437
Title: Non Interventional Study in Slovak Patients With Primary Open Angle Glaucoma and/or Ocular Hypertension Treated With Xalacom® After Failure of Previous Antiglaucoma Therapy Due to Ineffectivity or Intolerance.
Brief Title: Non Interventional Study With Primary Open Angle Glaucoma and/or Ocular Hypertension Patients Treated With Xalacom® After Failure of Previous Antiglaucoma Therapy.
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6641053
Record Dates: First submitted 2008-11-19; First posted 2008-12-03 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2011-06

CONDITIONS: Glaucoma, Open-angle
Keywords: glaucoma, open-angle, non-interventional study, safety, tolerability
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Xalacom

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Xalacom treatment: patients with primary glaucoma
  Interventions: Drug: Xalacom

INTERVENTIONS:
Drug: Xalacom — Xalacom 1 drop into the affected eye daily

SUMMARY:
This study is designed to evaluate the safety and tolerability of Xalacom in patients with primary glaucoma

DETAILED DESCRIPTION:
according to physicians decision, patients who met inclusion and exclusion criteria and sign the ICD

ELIGIBILITY:
Inclusion Criteria:

* primary open angle glaucoma
* ocular hypertension
* age >18 years

Exclusion Criteria:

* bradycardia
* obstructive pulmonary disease
* hypersensitivity to the drug

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years with primary open angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular hyperemia | 12 months
safety of treatment | 12 months

SECONDARY OUTCOMES:
effectiveness in IOP lowering | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- Slovakia (35):
  - Pfizer Investigational Site, Banovce N. Bebravou
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bojnice
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Brezno
  - Pfizer Investigational Site, Dunajská Streda
  - Pfizer Investigational Site, Galanta
  - Pfizer Investigational Site, Kežmarok
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Krompachy
  - Pfizer Investigational Site, Lipany
  - Pfizer Investigational Site, Lučenec
  - Pfizer Investigational Site, Martin
  - Pfizer Investigational Site, Myjava
  - Pfizer Investigational Site, Nitra
  - Pfizer Investigational Site, Nová Baňa
  - Pfizer Investigational Site, Nove Mesto N. Vahom
  - Pfizer Investigational Site, Nové Zámky
  - Pfizer Investigational Site, Poprad
  - Pfizer Investigational Site, Prešov
  - Pfizer Investigational Site, Rimavská Sobota
  - Pfizer Investigational Site, Rožňava
  - Pfizer Investigational Site, Ružomberok
  - Pfizer Investigational Site, Sabinov
  - Pfizer Investigational Site, Sliač
  - Pfizer Investigational Site, Snina
  - Pfizer Investigational Site, Spišská Nová Ves
  - Pfizer Investigational Site, Stará Ľubovňa
  - Pfizer Investigational Site, Stará Turá
  - Pfizer Investigational Site, Šaľa
  - Pfizer Investigational Site, Topoľčany
  - Pfizer Investigational Site, Zlaté Moravce
  - Pfizer Investigational Site, Zvolen
  - Pfizer Investigational Site, Žiar nad Hronom
  - Pfizer Investigational Site, Žilina

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6641053&StudyName=Non%20interventional%20study%20with%20Primary%20Open%20Angle%20Glaucoma%20and/or%20Ocular%20Hypertension%20patients%20treated%20with%20Xalacom%AE%20after%20failure%20of%20pre